CLINICAL TRIAL: NCT00589238
Title: Randomised Phase II Trial of Neoadjuvant Weekly Paclitaxel Plus Carboplatin Compared to Weekly Paclitaxel Alone Followed in Both Arms by Doxorubicin and Cyclophosphamide for Operable or Locally Advanced Basal-like Subtype Breast Cancer Correlating BRCA-1 mRNA and Protein Expression With Carboplatin Response
Brief Title: Paclitaxel, Doxorubicin, and Cyclophosphamide With Or Without Carboplatin in Treating Women With Locally Advanced Breast Cancer That Can Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Yap Yoon Sim, Senior Consultant, National Cancer Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000579522; SINGAPORE-NCC-0701
Record Dates: First submitted 2008-01-03; First posted 2008-01-09 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Paclitaxel

ARMS (2):
- Arm 1 (Standard Arm) (Other): Arm 1 (Standard Arm) Preoperative (primary/ neoadjuvant) intravenous weekly paclitaxel 80 mg/m2 for 12 weeks followed by doxorubicin 60 mg/m2 in combination with cyclophosphamide 600 mg/m2 every 21 days for 4 cycles.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Arm 2 (Experimental Arm) (Experimental): Arm 2 (Experimental Arm) Preoperative intravenous weekly paclitaxel 80 mg/m2 in combination with carboplatin AUC 2 on D1, D8 and D15 every 28 days for 4 cycles followed by doxorubicin 60 mg/m2 in combination with cyclophosphamide 600 mg/m2 every 21 days for 4 cycles.
  Interventions: Drug: carboplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
  Arms: Arm 2 (Experimental Arm)
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, doxorubicin, cyclophosphamide, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether combination chemotherapy is more effective with or without carboplatin in treating breast cancer.

PURPOSE: This randomized phase II trial is studying giving paclitaxel together with doxorubicin and cyclophosphamide to see how well it works compared to giving paclitaxel together with doxorubicin, cyclophosphamide, and carboplatin in treating women with locally advanced breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate tumor pathological complete response rate after neoadjuvant paclitaxel with vs without carboplatin followed by cyclophosphamide and doxorubicin hydrochloride in women with basal-type subtype primary breast cancer.

Secondary

* To evaluate the clinical and pathological overall response rate.
* To evaluate safety and toxicity.
* To evaluate disease-free survival and overall survival.
* To correlate low BRCA1 expression (protein and mRNA), p53 mutation, positive CK5/6, positive CK 14, basal-like gene expression profile, and response to carboplatin-based treatment.

OUTLINE: This is a multicenter study. Patients are stratified according to clinical stage (T2-3 vs T4). Patients are randomized to 1 of 2 treatment arms.

* Arm I (standard therapy): Patients receive paclitaxel IV over 1 hour once weekly in weeks 1-12. Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV on days 1, 8, and 15. Treatment with doxorubicin hydrochloride and cyclophosphamide repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (experimental therapy): Patients receive paclitaxel IV over 1 hour and carboplatin IV over 15 to 20 minutes on days 1, 8, and 15. Treatment with paclitaxel and carboplatin repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive doxorubicin hydrochloride and cyclophosphamide as in arm I.

All patients will then undergo surgical resection of the tumor.

Patients undergo biopsy for correlative studies. Samples are analyzed for estrogen receptor and progesterone receptor status, and molecular endpoints (CK 5/6, CK14, p53, BRCA, and EGFR) by RT-PCR, immunohistochemistry, protein expression, and gene expression profiling.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive basal-type breast cancer meeting the following criteria:

  * Newly diagnosed disease
  * Locally advanced or operable primary disease > 2 cm, without evidence of metastatic disease
  * Clinical T2 (> 2 cm), T3 (> 5 cm), or T4 primary tumors with or without clinical lymph node involvement (N0-3)

    * T4 tumors are defined by any of the following:

      * Skin ulceration
      * Satellite nodules
      * Peau d' orange (skin edema)
      * Chest wall invasion
      * Inflammatory breast cancer
* Her-2/neu 0-1+ by IHC (or negative by fluorescent in situ hybridization if Her-2 2+ by immunohistochemistry)
* No metastatic disease
* Hormone receptor status:

  * Estrogen and progesterone receptor-negative disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Female
* Menopausal status not specified
* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy > 10 years
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Cardiac ejection fraction ≥ 50% as assessed by MUGA scan or 2D echocardiogram

Exclusion criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel, carboplatin, or other agents used in the study
* Pre-existing peripheral neuropathy
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* Prior malignancies except for basal cell carcinoma of the skin or curatively treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No HIV-positive patients receiving combination antiretroviral therapy
* No concurrent primary growth factor prophylaxis
* No other concurrent investigational agents
* No other concurrent chemotherapy, immunotherapy, hormonal cancer therapy, surgery for cancer, or experimental medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pathological complete response rate | Pathological response will be assessed by evaluation of surgical specimen after completion of protocol treatment.

SECONDARY OUTCOMES:
Clinical and pathological overall response rates | Clinical response: Serial 4 weekly clinical examination; Mammography, breast ultrasound: Baseline, 3 weeks after treatment protocol or documented clinical progression. Pathological response: Evaluation of surgical specimen after protocol treatment.
Overall and disease-free survival | Clinical response: Serial 4 weekly clinical examination; Mammography, breast ultrasound: Baseline, 3 weeks after treatment protocol or documented clinical progression. Pathological response: Evaluation of surgical specimen after protocol treatment.
Incidence of each toxicity item | Clinical response: Serial 4 weekly clinical examination; Mammography, breast ultrasound: Baseline, 3 weeks after treatment protocol or documented clinical progression. Pathological response: Evaluation of surgical specimen after protocol treatment.
Correlation between low BRCA1 expression (protein and mRNA), p53 mutation, positive CK5/6, positive CK14, basal like gene expression profile, and response to carboplatin based treatment | Clinical response: Serial 4 weekly clinical examination; Mammography, breast ultrasound: Baseline, 3 weeks after treatment protocol or documented clinical progression. Pathological response: Evaluation of surgical specimen after protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wong Nan Soon, MBBS, MRCP, FAMS, Principal Investigator — National Cancer Centre, Singapore; Ann Lee Siew Gek, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre - Singapore, Singapore
  - KK Women's and Children Hospital, Singapore